CLINICAL TRIAL: NCT06352463
Title: More Than the Sum of Its Parts: Investigating a Combined Parent-child Treatment for Children With Social Anxiety
Brief Title: Intervention Social Anxiety: Combining Parent-child Treatment
Acronym: ISA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University (Other)
Collaborators: Leids Universitair Behandel en Expertise Centrum (LUBEC) (Unknown); GGZ Delfland (Unknown); Netherlands Organisation for Scientific Research (Other Government)
Responsible Party: Principal Investigator, Anke M Klein, AS, Principal Investigator, Leiden University
Organization: Leiden University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 406.XS.03.068
Record Dates: First submitted 2024-03-26; First posted 2024-04-08 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Social Anxiety Disorder of Childhood
MeSH Terms: interventions — Dichlorodiphenyldichloroethane

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 2-week waiting period (Active Comparator): Children and parents have to wait 2 weeks between baseline 1 and the start of the treatment. In the first week, they fill in ESMs daily.
  Interventions: Other: Denken + Doen = Durven; Other: Supportive Parenting for Anxious Childhood Emotions
- 4-week waiting period (Active Comparator): Children and parents have to wait 4 weeks between baseline 1 and the start of the treatment. In the first and third week, they fill in ESMs daily.
  Interventions: Other: Denken + Doen = Durven; Other: Supportive Parenting for Anxious Childhood Emotions
- 6-week waiting period (Active Comparator): Children and parents have to wait 6 weeks between baseline 1 and the start of the treatment. In the first, third, and fifth week, they fill in ESMs daily.
  Interventions: Other: Denken + Doen = Durven; Other: Supportive Parenting for Anxious Childhood Emotions

INTERVENTIONS:
Other: Denken + Doen = Durven — DDD is an evidence based cognitive behavioural therapy (CBT)-treatment protocol for children with anxiety. This research will use the modular version of DDD, which means that the therapist will decide which modules she will use based on the specific symptoms and needs of the child. DDD consists of four parts. First, there will be psycho education in which the child learns about how anxiety can arise, when anxiety is normal, and how thoughts, emotions, and behaviour are linked. Second, the child will learn coping strategies for dealing with anxiety. Third, there will be cognitive restructuring by which that the child will learn skills to deal with anxious and negative thoughts, through challenging and experimenting. Finally, there will be exposure. In the exposure sessions, the child will face their fears step by step.
  Other Names: DDD
Other: Supportive Parenting for Anxious Childhood Emotions — Parents will follow the SPACE program. SPACE is a theory driven, evidence-based treatment program of 12 sessions. In a structured way, parents are trained to change their own behaviour as a reaction to the symptoms of their child. First, they are trained to recognise family accommodation and slowly reduce this. Second, this program focuses on the increase in supportive reactions from parents. They are taught to accept the child's feelings, fears, and problems and to trust in the ability of the child to cope with and tolerate anxiety-related problems. These two goals are attained via a sequence of steps in the SPACE manual. Furthermore, SPACE includes additional modules that can be implemented if needed. These provide tools for conquering communal challenges that can arise during the treatment process, including dealing with extremely disruptive behaviour of children and improving parental collaboration.
  Other Names: SPACE

SUMMARY:
The aim of this pilot project is to investigate a treatment program for children with social anxiety, in which children and their parents, parallel to each other, follow separate evidence-based interventions. The added value of this pilot project is that the investigators are examining how both programs interact when offered simultaneously.

DETAILED DESCRIPTION:
After a diagnostic trajectory and a 2-week reflection period, children and their parents are invited to come into the lab for baseline 1. During baseline 1, children and their parents will be interviewed and they will fill in some questionnaires. They will then be randomly assigned to a 2-, 4-, or 6-week waiting period. During this waiting period they will fill in Experience Sampling Method (ESMs) daily, every other week. One week before the end of the waiting period, baseline 2 will take place. After the waiting period children and their parents will start their separate treatments in parallel. Children will get an individually tailored cognitive behavioural therapy (CBT)-protocol for social anxiety and parents will get SPACE. In the treatment period, they will fill in ESMs daily. There is another assessment with interviews and questionnaires at mid-treatment (after 6 sessions) and post-treatment (after 12 sessions), as well as 1- and 2-months after treatment has ended. After the treatment period, the frequency of the ESMs will go back to daily every other week.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis social anxiety
* At least 1 parent is willing to participate

Exclusion Criteria:

* Currently under treatment for anxiety
* Other complaints that need attention first
* Not understanding instructions/treatment

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in severity of social anxiety in children | From baseline to the end of treatment and follow-up (1 and 2 months post-treatment)
  Severity of social anxiety will be assessed using the Anxiety Disorder Interview Schedule (ADIS-V), which will provide a clinician severity rating (CSR)-score. This is a score between 0 and 8, with higher scores indicating a higher severity and interference of anxiety. The ADIS-V will be administered to children and parents.

SECONDARY OUTCOMES:
Change in anxiety-related symptoms and family accommodation | From baseline to the end of treatment and follow-up (1 and 2 months post-treatment)
  Children and their parents will fill in a daily experience sampling method (ESM) on their phone to measure thoughts, emotions, and behaviours in the flow of daily life. Children are asked 3 questions, each on a scale from 0 to 8. This sums up to a score between 0 and 24 each day for children. Parents are asked 7 questions which they answer on a scale between 0 and 4, resulting in a score between 0 and 28 each day for parents. Higher scores indicate more anxiety-related symptoms and family accommodation.

CONTACTS AND LOCATIONS:
Overall Officials: Anke M Klein, AS, Principal Investigator — Leiden University
Locations (3):
- Netherlands (3):
  - GGZ Delfland, Delft, South Holland
  - Leiden University, Leiden, South Holland
  - LUBEC, Leiden, South Holland

IPD SHARING:
Plan to Share IPD: No
The investigators will share the data upon request, but only for specific purposes. In addition, the data needs to be deleted after use. The investigators will not share data that cannot be anonymised, such as the video data.

REFERENCES:
- [Background] First MB. Diagnostic and statistical manual of mental disorders, 5th edition, and clinical utility. J Nerv Ment Dis. 2013 Sep;201(9):727-9. doi: 10.1097/NMD.0b013e3182a2168a. No abstract available. PMID 23995026
- [Background] Bulte I, Onghena P. Randomization tests for multiple-baseline designs: an extension of the SCRT-R package. Behav Res Methods. 2009 May;41(2):477-85. doi: 10.3758/BRM.41.2.477. PMID 19363188
- [Background] Craske MG, Treanor M, Zbozinek TD, Vervliet B. Optimizing exposure therapy with an inhibitory retrieval approach and the OptEx Nexus. Behav Res Ther. 2022 May;152:104069. doi: 10.1016/j.brat.2022.104069. Epub 2022 Mar 15. PMID 35325683
- [Background] Kagan ER, Peterman JS, Carper MM, Kendall PC. ACCOMMODATION AND TREATMENT OF ANXIOUS YOUTH. Depress Anxiety. 2016 Sep;33(9):840-7. doi: 10.1002/da.22520. Epub 2016 May 23. PMID 27213722
- [Background] Kazdin AE. Single-case experimental designs. Evaluating interventions in research and clinical practice. Behav Res Ther. 2019 Jun;117:3-17. doi: 10.1016/j.brat.2018.11.015. Epub 2018 Dec 2. PMID 30527785
- [Background] Krasny-Pacini A, Evans J. Single-case experimental designs to assess intervention effectiveness in rehabilitation: A practical guide. Ann Phys Rehabil Med. 2018 May;61(3):164-179. doi: 10.1016/j.rehab.2017.12.002. Epub 2017 Dec 15. PMID 29253607
- [Background] Lebowitz ER, Woolston J, Bar-Haim Y, Calvocoressi L, Dauser C, Warnick E, Scahill L, Chakir AR, Shechner T, Hermes H, Vitulano LA, King RA, Leckman JF. Family accommodation in pediatric anxiety disorders. Depress Anxiety. 2013 Jan;30(1):47-54. doi: 10.1002/da.21998. Epub 2012 Sep 10. PMID 22965863
- [Background] Lebowitz ER, Marin C, Martino A, Shimshoni Y, Silverman WK. Parent-Based Treatment as Efficacious as Cognitive-Behavioral Therapy for Childhood Anxiety: A Randomized Noninferiority Study of Supportive Parenting for Anxious Childhood Emotions. J Am Acad Child Adolesc Psychiatry. 2020 Mar;59(3):362-372. doi: 10.1016/j.jaac.2019.02.014. Epub 2019 Mar 7. PMID 30851397
- [Background] Norman KR, Silverman WK, Lebowitz ER. Family Accommodation of Child and Adolescent Anxiety: Mechanisms, Assessment, and Treatment. J Child Adolesc Psychiatr Nurs. 2015 Aug;28(3):131-40. doi: 10.1111/jcap.12116. Epub 2015 Aug 4. PMID 26238937
- [Background] Rapee RM, McLellan LF, Carl T, Trompeter N, Hudson JL, Jones MP, Wuthrich VM. Comparison of Transdiagnostic Treatment and Specialized Social Anxiety Treatment for Children and Adolescents With Social Anxiety Disorder: A Randomized Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2023 Jun;62(6):646-655. doi: 10.1016/j.jaac.2022.08.003. Epub 2022 Aug 17. PMID 35987298
- [Background] Scaini S, Belotti R, Ogliari A, Battaglia M. A comprehensive meta-analysis of cognitive-behavioral interventions for social anxiety disorder in children and adolescents. J Anxiety Disord. 2016 Aug;42:105-12. doi: 10.1016/j.janxdis.2016.05.008. Epub 2016 Jun 25. PMID 27399932
- [Background] Spence SH, Rapee RM. The etiology of social anxiety disorder: An evidence-based model. Behav Res Ther. 2016 Nov;86:50-67. doi: 10.1016/j.brat.2016.06.007. Epub 2016 Jul 1. PMID 27406470
- [Background] Force, T. (1995). Task Force on Promotion and Dissemination of Psychological Procedures. Training in and dissemination of empirically-validated treatments: report and recommendations. The Clinical Psychologist, 48(1), 3-23.
- [Background] Albano, A. M. & Silverman, W. K. (2022). Anxiety and related disorders interview schedule for DSM-5 (ADIS-5-PV). Oxford University Press, USA.
- [Background] van Steensel (2023). Database effective youth interventions: description 'Denken + Doen = Durven'. Utrecht: Nederlands Jeugdinstituut. Downloaded from www.nji.nl/jeugdinterventies.